CLINICAL TRIAL: NCT00634283
Title: Physiologic Monitoring of Antidepressant Medication Effects in Normal Healthy Subjects II
Brief Title: Study of the Effects of an Antidepressant Medication and Placebo on the Brain Functioning of Normal Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 07-10-051
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Subjects are assigned to one of two groups (antidepressant-experienced and antidepressant-naive) and receive parallel treatment (1 week of placebo followed by 4 weeks of venlafaxine) for the duration of the study. Subjects and assessors were blinded to treatment condition.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: We compared EEG outcomes for those subjects who had been randomly assigned to blinded treatment with venlafaxine (antidepressant-experienced, n=2) vs. placebo (antidepressant-naive, n=4). All subjects received 1 week of placebo followed by 4 weeks of venlafaxine. Subjects were blinded to the treatment during both phases of the study using lookalike capsules. Outcomes assessors and the treating physician also were blinded to treatment condition.
Oversight: Data Monitoring Committee: No

ARMS (2):
- antidepressant-experienced (Experimental): Subjects who had previously been exposed to active antidepressant medication (venlafaxine)
  Interventions: Drug: venlafaxine
- antidepressant-naive (Placebo Comparator): Subjects who had previously been exposed to placebo only (and never to active antidepressant medication)
  Interventions: Drug: venlafaxine

INTERVENTIONS:
Drug: venlafaxine — venlafaxine IR 150mg
  Other Names: Effexor

SUMMARY:
This study examines the effects of an antidepressant medication and placebo on the brain functioning of normal subjects. In this study, recordings of brain electrical activity are being used to detect and monitor the response to treatment with venlafaxine IR (Effexor), a drug used for the treatment of depression. The intent of this study is to test specific hypotheses regarding:

1. long-term brain effects of a single course of antidepressant treatment
2. pharmaco-conditioning effects underlying antidepressant tolerance/sensitization
3. brain functional response to initial versus subsequent antidepressant trials in normal healthy subjects.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a lifelong and recurrent illness, such that many individuals require multiple courses of antidepressant medication treatment. While some patients respond completely to each course of treatment, many do not, and with each unsuccessful antidepressant trial the likelihood that a patient will respond decreases. This raises the possibility that neurophysiologic response in subsequent antidepressant treatment may be influenced by learning processes including sensitization, habituation, and/or classical conditioning. Classical conditioning would entail the association of cues such as pill-taking (conditioned stimuli; CS) with the effects of active medication (unconditioned stimulus; US), such that later presentation of the CS alone would come to elicit a conditioned response (CR). Such effects could be revealed by blinded administration of placebo following a period of treatment with active medication. Habituation effects (tolerance), or sensitization effects (increased response), which require only repeated exposure to a stimulus, might be evidenced after repeated courses of antidepressant treatment. Knowledge of how learning processes impact neurophysiologic response to successive courses of antidepressant treatment would have relevance for clinical populations. Specific hypotheses, however, may be tested in healthy non-clinical samples to avoid potential confounding factors related to severity or chronicity of illness. Learning theories would suggest two hypotheses: (1) neurophysiologic response to placebo will differ between subjects who were previously treated with antidepressant treatment as compared to placebo (classical conditioning hypothesis); and (2) neurophysiologic response to an initial course of antidepressant treatment will differ from response to a repeated course of antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject age is 18-75 years
* Subject must be in overall good health (i.e., free of any medical condition known to affect brain function).
* Subject must have participated in former study, Physiologic Monitoring of Antidepressant Medication Effects in Normal Controls Subjects (IRB#: 00-11-038-13)
* Subject has had a normal physical exam within one year prior to entry of the study
* Capacity to give Informed Consent

Exclusion Criteria:

* Subject has serious medical illness, such as high blood pressure, heart disease, renal impairment, or cirrhosis of the liver.
* Subject meets DSM-IV Axis I criteria for a mood, anxiety, cognitive, or psychiatric disorder; or meets criteria for cluster A or B axis II diagnoses. These disorders will be determined on the basis of a structured assessment with the MINI (Mini International Neuropsychiatric Interview for DSM-IV Axis I Disorders)
* Subject has a history of current or past active suicidal ideation or suicide attempts.
* Subject has received treatment with an antidepressant medication or any medications that could influence brain function since his/her participation in the initial study
* Subject is using any of the following medications which interfere with EEG measures of brain function: Anticholinergics, Barbiturates, Benzodiazepines, Sedating Antihistamines (e.g. diphenhydramine (Benadryl) would be exclusionary, but not loratadine (Claritin))
* Subject has a history of seizures, brain surgery, skull fracture, significant head trauma, or previous abnormal EEG
* Subject is pregnant or planning on becoming pregnancy during course of the study
* Subject is a UCLA student or staff member directly under instruction or employment of any of the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Leuchter, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles (UCLA), Los Angeles, California, United States

REFERENCES:
- [Result] Hunter AM, Cook IA, Abrams M, Leuchter AF. Neurophysiologic effects of repeated exposure to antidepressant medication: are brain functional changes during antidepressant administration influenced by learning processes? Med Hypotheses. 2013 Dec;81(6):1004-11. doi: 10.1016/j.mehy.2013.09.016. Epub 2013 Sep 17. PMID 24112999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 142 research subjects were enrolled at the Laboratory of Brain, Behavior and Pharmacology from 8/19/05-9/30/08.
Pre-assignment Details: Subjects were required to wash out from any exclusionary medication for at least two weeks. Subjects taking fluoxetine were required to wash out for at least 30 days prior to treatment assignment.
Groups:
- Venlafaxine IR (Effexor): Five weeks of treatment with venlafaxine IR
Period: Overall Study
Arm/Group | Venlafaxine IR (Effexor)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Venlafaxine IR (Effexor)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — 18 years to 65 years of age. Must be in good health (i.e., free of any medical condition known to affect brain function).
  years | 46.5 (1)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants must be 18-75 years old, in overall good health, must have participated in the former study Physiologic Monitoring of Antidepressant Medication Effects in Normal Controls Subjects, has had a normal physical exam one year prior to entry of the study, has the capacity to give informed consent.
  Participants
    Female | 6
    Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Changes in Quantitative Electroencephalogram (qEEG) Prefrontal Cordance (PFC) Over Time (4 Weeks).
Description: Cordance values were calculated from conventional 'absolute' and 'relative' qEEG power measures using a three-step procedure. First, EEG power values were computed using a re-attributional electrode montage. Second, the absolute and relative power values were z-transformed to measure deviation from the mean values for each electrode site s in each frequency band f for that recording, yielding Anorm(s,f) and Rnorm(s,f), respectively. Third, these z-scores were summed to yield a cordance "intensity" value, Z, for each electrode in each frequency band where Z(s,f) = Anorm(s,f) + Rnorm(s,f). Analyses for this report focused on changes-from-baseline theta-band (8-12Hz) cordance in the prefrontal region (electrodes Fp1, Fpz, Fp2). Results are defined in terms of positive and negative change where a positive change represents an increased physiologic and behavioral response to the drug (sensitization) and a negative change represents an increased tolerance to the drug (habituation).
Time Frame: Average over 4 weeks
Population: Antidepressant-experienced subjects; n=2 and antidepressant-naive subjects; n=4
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Antidepressant Treatment-experienced: Subjects in this group had prior exposures to antidepressant medication (venlafaxine)
- Antidepressant Treatment-naive: Subjects in this group had never before been exposed to antidepressant medication
Arm/Group | Antidepressant Treatment-experienced | Antidepressant Treatment-naive
Number analyzed (Participants) | 2 | 4
z-score
  PFC change after placebo lead-in | -0.54 (0.44) | -0.09 (0.46)
  PFC at Baseline | -0.09 (0.86) | -0.88 (1.55)
Statistical Analysis 1: Comparison: Antidepressant Treatment-experienced vs Antidepressant Treatment-naive; Test type: Superiority; p = 0.55, t-test, 2 sided
Statistical Analysis 2: Comparison: Antidepressant Treatment-experienced vs Antidepressant Treatment-naive; Change in PFC over the one-week placebo lead-in period was compared between antidepressant-experienced and antidepressant-naive groups using a between groups t-test; Test type: Superiority; p = 0.32, t-test, 2 sided — The a priori threshold was set at 0.05, 2-tailed, without adjustment for multiple comparisons; Group differences in PFC changes over time during administration of venlafaxine were assessed using mixed-model analysis. we compared brain functional changes over the course of venlafaxine treatment between antidepressant-experienced and antidepressant-naïve subjects using linear mixed model analysis (random intercept model) conducted using full maximum likelihood estimation (MLE). Changes in PFC were calculated from the end of placebo lead-in to 48 hours, and 1, 2, and 4 weeks, yielding a within-group factor of time with four levels. We employed a first-order autoregressive covariance structure to reflect our assumption that PFC measurements closer together in time would be more highly correlated

2. Primary Outcome: Changes in Quantitative Electroencephalogram (qEEG) Prefrontal Cordance (PFC) Over 1 Week Placebo lead-in.
Description: as for outcome 1
Time Frame: 1-week placebo lead-in
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Antidepressant Treatment-experienced | Antidepressant Treatment-naive
Number analyzed (Participants) | 2 | 4
Z-score | -0.54 (0.44) | -0.09 (0.46)

ADVERSE EVENTS:
Groups:
- Antidepressant Treatment-experienced: Healthy subjects who have been previously exposed to venlafaxine
- Antidepressant Treatment-naive: Healthy subjects who have never been previously exposed to antidepressant medication
Arm/Group | Antidepressant Treatment-experienced | Antidepressant Treatment-naive
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No